CLINICAL TRIAL: NCT01811420
Title: Chemomechanical Caries Removal Using a Papain-Based Gel: A Randomized Clinical Trial
Brief Title: Chemomechanical Caries Removal Using Papain Gel
Acronym: CMCR09
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Lara Jansiski Motta, PhD Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cariesremoval09
Record Dates: First submitted 2013-03-06; First posted 2013-03-14 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Dental Caries
Keywords: dental caries; caries removal; chemomechanical caries removal
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHEMOMECHANICAL CARIES REMOVAL (Experimental): Dental caries removal using papain based gel
  Interventions: Procedure: Chemomechanical Caries Removal
- conventional method (Active Comparator): Dental caries removal using rotatory instrument
  Interventions: Procedure: Conventional method

INTERVENTIONS:
Procedure: Chemomechanical Caries Removal — Chemomechanical Caries Removal Using A Papain-Based Gel
  Arms: CHEMOMECHANICAL CARIES REMOVAL
Procedure: Conventional method — Dental caries removal using rotatory instrument
  Arms: conventional method

SUMMARY:
To evaluate the efficacy of a papain-based gel in caries removal.

DETAILED DESCRIPTION:
Twenty children with at least two carious molar teeth without pulpal involvement participated in this randomized clinical trial. A total of 40 teeth were randomly divided into two treatment groups: group A, papain-based gel; and group B, conventional technique. Data collection included the time required for caries removal, need for local anesthesia, degree of discomfort, changes in the number of viable bacteria, and clinical evaluation of glass ionomer-cement restorations 6-month post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children with active caries without pulpal involvement in two deciduous molar teeth participated in the trial.
* The caries were located on the occlusal surface.

Exclusion Criteria:

* Children with pathological process of the dental tissue, with pulpal involvement

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
restauration evaluation | 18 months
  the restauration will be assessed by clinical examination for detection the current caries

SECONDARY OUTCOMES:
discomfort or pain | 6 months
  The Faces Pain Scale was used to evaluate the need for local anesthesia during the procedure. The child was asked to choose a face matching the intensity of his or her pain experience during the procedure.

OTHER OUTCOMES:
radiographic status | 18 months
  the restauration will be assessed by radiographic examination for detection the current caries

CONTACTS AND LOCATIONS:
Overall Officials: Lara J Motta, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- Universidade Nove de Julho, São Paulo, Sao Apaulo, Brazil

REFERENCES:
- [Derived] Motta LJ, Bussadori SK, Campanelli AP, Silva AL, Alfaya TA, Godoy CH, Navarro MF. Efficacy of Papacarie((R)) in reduction of residual bacteria in deciduous teeth: a randomized, controlled clinical trial. Clinics (Sao Paulo). 2014;69(5):319-22. doi: 10.6061/clinics/2014(05)04. PMID 24838896
- [Derived] Motta LJ, Bussadori SK, Campanelli AP, da Silva AL, Alfaya TA, de Godoy CH, Navarro MF. Pain during Removal of Carious Lesions in Children: A Randomized Controlled Clinical Trial. Int J Dent. 2013;2013:896381. doi: 10.1155/2013/896381. Epub 2013 Dec 4. PMID 24363672